CLINICAL TRIAL: NCT02111083
Title: Evaluation of the Bioequivalence of Two Formulations of Insulin Lispro in Healthy Subjects
Brief Title: A Study of 2 Different Formulations of Insulin Lispro in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 15418; F3Z-EW-IOQM (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Lispro A (Active Comparator): Insulin Lispro A 20 units (U) of strength 200 units per milliliter (U/mL) (U-200)administered subcutaneously (SC) once in two of four study periods.(Two doses of test [T]).
  Interventions: Biological: Insulin Lispro
- Insulin Lispro B (Experimental): Insulin Lispro B 20 units (U) of strength 100 U/mL (U-100) administered SC once in two of four study periods.(Two doses of reference [R]).
  Interventions: Biological: Insulin Lispro

INTERVENTIONS:
Biological: Insulin Lispro — LY275585 administered SC.

SUMMARY:
The study involves 4 injections of insulin lispro and its purpose is to:

* Determine if 2 formulations of insulin lispro are treated by the body in a similar way.
* Compare how the 2 formulations of insulin lispro affect blood sugar level.
* Determine the safety of each insulin lispro formulations and any side effects that might be associated with them when given to healthy participants. The study is expected to last up to approximately 9 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Are healthy males or females
* Body mass index (BMI) between 18.5 and 29.9 kilogram per meter squared (kg/m^2)
* Are nonsmokers
* Have normal blood pressure and pulse rate, a normal electrocardiogram (ECG), and clinical laboratory test results within normal reference range at screening.

Exclusion Criteria:

* History of first-degree relatives known to have diabetes mellitus
* Evidence of significant active neuropsychiatric disease
* Evidence of an acute infection with fever or infectious disease
* Intend to use over-the-counter or prescription medication (apart from vitamin/mineral supplements, occasional paracetamol, or birth control methods).
* Have used systemic glucocorticoids within 3 months prior to entry into the study.
* Have donated blood of 1 unit or more within the last 3 months prior to study entry
* Excessive alcohol intake
* Have a fasting venous blood glucose (fasting blood glucose [FBG], plasma) >6 millimoles per liter (mmol/L) at screening
* Have positive hepatitis B surface antigen.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Lispro Dosing Sequence TRTR: Each subject was administered insulin lispro A 20 units (U) of strength 200 units per milliliter (U/mL) (U-200) (test [T] on 2 occasions) and insulin lispro B 20 units (U) of strength 100 U/mL (U-100) (reference [R] on 2 occasions).Subjects were randomly assigned to dosing sequences TRTR.
- Insulin Lispro Dosing Sequence RTRT: Each subject was administered insulin lispro A 20 units (U) of strength 200 units per milliliter (U/mL) (U-200) (test [T] on 2 occasions) and insulin lispro B 20 units (U) of strength 100 U/mL (U-100) (reference [R] on 2 occasions).Subjects were randomly assigned to dosing sequences RTRT.
Period: First Intervention (1 Day)
Arm/Group | Insulin Lispro Dosing Sequence TRTR | Insulin Lispro Dosing Sequence RTRT
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Interval Between Dosing (7-8 Days)
Arm/Group | Insulin Lispro Dosing Sequence TRTR | Insulin Lispro Dosing Sequence RTRT
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Insulin Lispro Dosing Sequence TRTR | Insulin Lispro Dosing Sequence RTRT
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Interval Between Dosing (7-8 Days)
Arm/Group | Insulin Lispro Dosing Sequence TRTR | Insulin Lispro Dosing Sequence RTRT
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | Insulin Lispro Dosing Sequence TRTR | Insulin Lispro Dosing Sequence RTRT
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Interval Between Dosing (7-8 Days)
Arm/Group | Insulin Lispro Dosing Sequence TRTR | Insulin Lispro Dosing Sequence RTRT
Started | 19 | 19
Completed | 18 | 18
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1
Period: Fourth Intervention (1 Day)
Arm/Group | Insulin Lispro Dosing Sequence TRTR | Insulin Lispro Dosing Sequence RTRT
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Insulin Lispro Dosing Sequence TRTR: Each subject was administered insulin lispro A U-200 (test [T] on 2 occasions) and insulin lispro B U-100(reference [R] on 2 occasions).Subjects were randomly assigned to dosing sequences TRTR.
- Insulin Lispro Dosing Sequence RTRT: Each subject was administered insulin lispro A U-200 (test [T] on 2 occasions) and insulin lispro B U-100 (reference [R] on 2 occasions). Subjects were randomly assigned to dosing sequences RTRT.
- Total: Total of all reporting groups
Arm/Group | Insulin Lispro Dosing Sequence TRTR | Insulin Lispro Dosing Sequence RTRT | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (6.1) | 30.4 (8.2) | 31.7 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 17 | 18 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameter: Area Under the Serum Insulin Concentration Versus Time Curve From Zero to Time of Return to Baseline (AUC0-tlast)
Time Frame: Day 1, predose through 8 hours post dose in each period.
Population: All participants who had at least one study treatment and had evaluable pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole*hour/liter (pmol*h/L)
Groups:
- Insulin Lispro A: Insulin Lispro A U-200 administered subcutaneously (SC) once in two of four study periods. (Two doses of test [T]).
- Insulin Lispro B: Insulin Lispro B U-100 administered SC once in two of four study periods. (Two doses of reference [R]).
Arm/Group | Insulin Lispro A | Insulin Lispro B
Number analyzed (Participants) | 38 | 38
picomole*hour/liter (pmol*h/L) | 2200 (16) | 2230 (17)
Statistical Analysis 1: Comparison: Insulin Lispro A vs Insulin Lispro B; Test type: Superiority or Other; Ratio of geometric least square means = 0.986, 90% CI 2-sided [0.965 to 1.01]

2. Primary Outcome: Pharmacokinetic Parameter: Maximum Serum Insulin Concentration (Cmax)
Time Frame: Day 1, predose through 8 hours post dose in each period
Population: All participants who had at least one study treatment and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole/liter (pmol/L)
Arm/Group | Insulin Lispro A | Insulin Lispro B
Number analyzed (Participants) | 38 | 38
picomole/liter (pmol/L) | 744 (38) | 851 (38)
Statistical Analysis 1: Comparison: Insulin Lispro A vs Insulin Lispro B; Test type: Superiority or Other; Ratio of geometric least square means = 0.872, 90% CI 2-sided [0.828 to 0.919]

3. Secondary Outcome: Pharmacokinetic Parameter: Time of Maximum Observed Serum Concentration (Tmax)
Time Frame: Day 1, predose through 8 hours post dose in each period.
Population: All participants who had at least one study treatment and had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Insulin Lispro A | Insulin Lispro B
Number analyzed (Participants) | 38 | 38
hours | 1 [0.5 to 3.0] | 1 [0.5 to 2.0]
Statistical Analysis 1: Comparison: Insulin Lispro A vs Insulin Lispro B; Test type: Superiority or Other; Median Difference (Final Values) = 0.25, 90% CI 2-sided [0 to 0.375]

4. Secondary Outcome: Pharmacodynamic Parameter: Total Amount of Glucose Infused (Gtot)
Description: The total amount of glucose infused during the euglycemic clamp procedure.
Time Frame: Day1, predose through 8 hours post dose in each period.
Population: All participants who had at least one study treatment and had evaluable pharmacodynamic(PD) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: grams (g)
Arm/Group | Insulin Lispro A | Insulin Lispro B
Number analyzed (Participants) | 38 | 38
grams (g) | 120 (31) | 120 (33)
Statistical Analysis 1: Comparison: Insulin Lispro A vs Insulin Lispro B; Test type: Superiority or Other; Ratio of geometric least square means = 0.986, 90% CI 2-sided [0.954 to 1.02]

5. Secondary Outcome: Pharmacodynamic Parameter: Maximum Glucose Infusion Rate (Rmax)
Description: The maximum observed glucose infusion rate during the euglycemic clamp procedure.
Time Frame: Day 1, predose through 8 hours post dose in each period.
Population: All participants who had at least one study treatment and had evaluable PD data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per minute (mg/min)
Arm/Group | Insulin Lispro A | Insulin Lispro B
Number analyzed (Participants) | 38 | 38
milligrams per minute (mg/min) | 503 (36) | 526 (36)
Statistical Analysis 1: Comparison: Insulin Lispro A vs Insulin Lispro B; Test type: Superiority or Other; Ratio of geometric least square means = 0.950, 90% CI 2-sided [0.901 to 1.00]

6. Secondary Outcome: Pharmacodynamic Parameter: Time of Maximum Glucose Infusion Rate (tRmax)
Time Frame: Day 1, predose through 8 hours post dose in each period.
Population: All participants who had at least one study treatment and had evaluable PD data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Insulin Lispro A | Insulin Lispro B
Number analyzed (Participants) | 38 | 38
hours | 2.71 (52) | 2.32 (52)
Statistical Analysis 1: Comparison: Insulin Lispro A vs Insulin Lispro B; Test type: Superiority or Other; Difference of least squares means = 0.424, 90% CI 2-sided [0.164 to 0.685]

7. Primary Outcome: Pharmacokinetic Parameter: Area Under the Curve(AUC)
Time Frame: Zero to infinity [AUC(0-∞)]
Population: All participants who had at least one study treatment and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole*hour/liter (pmol*h/L)
Arm/Group | Insulin Lispro A | Insulin Lispro B
Number analyzed (Participants) | 38 | 38
picomole*hour/liter (pmol*h/L) | 2330 (15) | 2360 (16)
Statistical Analysis 1: Comparison: Insulin Lispro A vs Insulin Lispro B; Test type: Superiority or Other; Ratio of geometric least square means = 0.992, 90% CI 2-sided [0.975 to 1.01]

ADVERSE EVENTS:
Groups:
- Insulin Lispro A: Insulin Lispro A U-200 subcutaneously (SC) once in two of four study periods. (Two doses of test [T]).
Arm/Group | Insulin Lispro A | Insulin Lispro B
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 21/38 | 16/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro A (N=38) | Insulin Lispro B (N=38)
Application site erythema (General disorders) | 2 (3) | 1 (2)
Catheter site related reaction (General disorders) | 7 (9) | 5 (5)
Infusion site bruising (General disorders) | 3 (3) | 1 (1)
Infusion site pain (General disorders) | 5 (5) | 4 (4)
Infusion site swelling (General disorders) | 5 (5) | 4 (5)
Injection site bruising (General disorders) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Vessel puncture site bruise (General disorders) | 1 (1) | 2 (2)
Vessel puncture site pain (General disorders) | 2 (2) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes